CLINICAL TRIAL: NCT03348319
Title: The Pancreas and the Bilio-pancreatic Junction: Is There a Pancreatic Segmentation Based on the Pancreatic Duct Branching?
Brief Title: Is There a Pancreatic Segmentation Based on the Pancreatic Duct Branching?
Status: Withdrawn | Type: Observational
Why Stopped: logistics problems
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA16146*
Record Dates: First submitted 2017-10-20; First posted 2017-11-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pancreas
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pancreas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cadaver organs
  Interventions: Other: radiation

INTERVENTIONS:
Other: radiation — Scanning cadaver organs

SUMMARY:
Limited pancreatic resections are increasingly performed, but the rate of postoperative fistula is higher than after classical resections. Pancreatic segmentation, anatomically and radiologically identifiable, may theoretically help the surgeon removing selected anatomical portions with their own segmental pancreatic duct and thus might decrease the postoperative fistula rate. Current pancreatic segmentation theories do not enable defining anatomical-surgical pancreatic segments. To our knowledge, no study has tried to describe pancreatic segmentation from the divisions of the pancreatic ducts to date. Hence, we hypothesize to explore the possibility of pancreatic segmentation following pancreatic ducts, using extensive reconstructions of pancreatic duct using micro-scanner on injected human pancreas.

DETAILED DESCRIPTION:
* In a first step, the injection technique will be developed (dilution, stability, hardening of the contrast mixture).
* In a second step, we will inject the mixture in human pancreas: into the duct tree, the vein and arteries. After hardening, the human pancreas will be removed from cadavers following the organ donation technique. The anatomic specimens will be scanned in the laboratory UMR CNRS 7369 MEDyC, Reims (Pr X. MAQUART, Dr J. DEVY).
* The images obtained (Dicom format) are very big in term of file size. Analysis of the images will be performed using a supercomputer of the laboratory CReSTIC - ROMEO EA 3804, Reims (Dr A. RENARD, Pr M. KRAJEKI). 3D reconstructions will be performed.

ELIGIBILITY:
inclusion criteria :

* All consecutive cadavers donated to the Department of Anatomy, Faculty of Medicine and University Hospital, Champagne-Ardenne University for anatomical education and research will be studied. These cadavers will be studied following all the ethical rules of work on cadaver material in our institution.

exclusion criteria :

* Cadavers not usable due to learning necessity, to failure of conservation, dissection difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive cadavers donated to the Department of Anatomy, Faculty of Medicine and University Hospital, Champagne-Ardenne University
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Size of the ducts | baseline
  The anatomic specimens will be scanned. The images will be analysed
Number of branching | baseline
  The anatomic specimens will be scanned. The images will be analysed